CLINICAL TRIAL: NCT03168386
Title: Effect of Intensive Motor Rehabilitation in Subacute Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, MD, PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-07-148
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Rehabilitation; Motor Function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Intenstive motor rehabilitation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive motor rehabilitation group (Experimental)
  Interventions: Procedure: Intensive motor rehabilitation

INTERVENTIONS:
Procedure: Intensive motor rehabilitation — Intensive motor rehabilitation during subacute stroke phase

SUMMARY:
Early stroke rehabilitation is known to be an effective and essential therapy in gaining functional independence and preventing complications. However, there was no consensus of proper amount of motor rehabilitation in stroke patients. In this study, the investigators investigated the effects of the intensive motor rehabilitation during subacute phase to improve motor function at 6 months after onset in patients with first-ever strokes.

DETAILED DESCRIPTION:
Intensive cognitive rehabilitation group

- physical and occupational therapy for 3 hours on every working day for 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* Acute first-ever stroke
* Upper limb score of Fugl-Meyer assessment at 7 days after onset : 25~84

Exclusion Criteria:

* Transient ischemic stroke
* Joint contracture of affected upper extremity

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Upper limb score of Fugl-Meyer assessment | Change of upper limb score of Fugl-Meyer assessment after intensive motor rehabilitation for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang WH, Sohn MK, Lee J, Kim DY, Lee SG, Shin YI, Oh GJ, Lee YS, Joo MC, Han EY, Kim YH. Korean Stroke Cohort for functioning and rehabilitation (KOSCO): study rationale and protocol of a multi-centre prospective cohort study. BMC Neurol. 2015 Mar 25;15:42. doi: 10.1186/s12883-015-0293-5. PMID 25886039